CLINICAL TRIAL: NCT05245877
Title: Pre- Vs. Postoperative Thromboprophylaxis in Pancreatic Surgery - a Prospective, Multicenter, Randomized Controlled Trial (PREPOSTEROUS Pancreas Trial)
Brief Title: Pre- Vs. Postoperative Thromboprophylaxis in Pancreatic Surgery
Acronym: PREPOSTEROUS2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, Primary investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HYKS-PREPOSTEROUS2
Record Dates: First submitted 2021-12-29; First posted 2022-02-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm; Surgery; Thrombosis; Bleeding
MeSH Terms: conditions — Pancreatic Neoplasms; Thrombosis; Hemorrhage | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative thromboprophylaxis (Experimental): Preoperatively initiated tromboprophylaxis
  Interventions: Drug: enoxaparin/tinzaparin/dalteparin
- Postoperative thromboprophylaxis (No Intervention): Postoperatively initiated thromboprophylaxis

INTERVENTIONS:
Drug: enoxaparin/tinzaparin/dalteparin — Patients randomized to the preoperative thromboprophylaxis will have their thromboprophylaxis initiated approximately 2-14 hours prior to the planned pancreatic surgery skin incision (depending on the center's current practice and logistics). Thromboprophylaxis can be initiated using enoxaparin (20 - 40 mg), tinzaparin (2500 - 4500 IU), or dalteparin (2500 - 5000 IU), with the dose based on patient's renal function according to the local standard of care. A center may reduce the dose 25-50% if the dose is given very close to the skin incision (i.e. at the morning of the operation instead of the evening before the operation).
  Arms: Preoperative thromboprophylaxis

SUMMARY:
Thromboprophylaxis for pancreatic surgery can be commenced either preoperatively or postoperatively. Despite a clear trade-off between thrombosis and bleeding in pancreatic surgery patients, there is no international consensus when thrombosis prophylaxis should be commenced in patients undergoing pancreatic surgery. There are no prospective randomized trials in this field, and current guidelines are unfortunately based on very low quality evidence, that is, a few retrospective studies and expert opinion. Both American and European thromboprophylaxis guidelines for abdominal cancer surgery support the preoperative initiation of thromboprophylaxis, but these guidelines do not specifically address the increased bleeding risk associated with pancreatic surgery. On the contrary, Dutch guidelines recommend postoperative thromboprophylaxis only, because of lack of evidence for preoperative thromboprophylaxis. Enhanced Recovery After Surgery (ERAS) Society Guidelines recommend preoperative thromboprophylaxis in pancreatic surgery, but the guidelines provide no supporting evidence for this recommendation. Overall, the amount of evidence is scarce and somewhat contradictory in this clinically relevant field of thromboprophylaxis in pancreatic surgery. The aim of this study is to compare pre- and postoperatively initiated thromboprophylaxis regimens in pancreatic surgery in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing either

1. pancreaticoduodenectomy or total pancreatectomy (for any indication) or
2. distal pancreatectomy for suspicion of cancer

Exclusion Criteria:

1. Patient on anticoagulative medication (heparin, low-molecular weight heparin, warfarin, direct oral anticoagulants) during the month (30 days) preceding surgery
2. Emergency operation (e.g. for trauma, infection or pancreatitis)
3. Age < 18 years
4. Allergy or other contraindication to planned low-molecular weight heparin
5. Inability to give written informed consent
6. Pancreatic resection not performed (removed from analyses after randomization)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism, number of patients | within 30 days from pancreatic resection
  Number of patients that have venous thromboembolism, which include any of the following: 1) symptomatic deep venous thromboembolism (including all deep veins e.g. all extremities, portal-, and superior mesenteric vein) diagnosed using ultrasound or computed tomography or magnetic resonance imaging, or in re-laparotomy/surgery, 2) pulmonary embolism diagnosed using computed tomography, magnetic resonance imaging, or lung perfusion imaging, or 3) death due to venous thromboembolism.

SECONDARY OUTCOMES:
Postpancreatectomy hemorrhage (PPH) | within 30 days from pancreatic resection
  Postpancreatectomy hemorrhage (PPH), any grade in ISGPS classification for postpancreatectomy hemorrhage, number of patients
Comprehensive Complication Index - score | within 30 days from pancreatic resection
  Comprehensive Complication Index - score
Length of postoperative hospital stay, | within 30 days from pancreatic resection
  Length of postoperative hospital stay, days, within 30 days from pancreas resection including hospital stay due to readmission(s)
Transfused red blood cells | during and within 30 days from pancreas resection
  Total amount of transfused red blood cells, units, during and within 30 days from pancreas resection
Post-operative hemoglobin below 70 g/l | during and within 30 days from pancreas resection
  Number of patients with post-operative hemoglobin below 70 g/l

CONTACTS AND LOCATIONS:
Locations (5):
- Sunnybrook Health Sciences Centre, Toronto, Canada
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided